CLINICAL TRIAL: NCT06154590
Title: Anastrozole Adjuvant Trial - Study of Anastrozole Compared to NOLVADEX (Tamoxifen Citrate) for Adjuvant Treatment of Early Breast Cancer (Clinical Studies), Tamoxifen Citrate Was Added to Adjunct Cytotoxic Chemotherapy- Treatment of Malignant Joint Tumor.
Brief Title: Anastrozole Adjuvant Trial - Study of Anastrozole Compared to NOLVADEX (Tamoxifen Citrate) for Adjuvant Treatment of Early Breast Cancer Clinical Studies), Adjunct Cytotoxic Chemotherapy and Malignant Joint Tumor
Acronym: NASBP-B-09
Status: Not yet recruiting | Type: Observational
Sponsor: DR. DIANE CHISESI NFS. MD. PHD. (Other)
Collaborators: IRB (Unknown)
Responsible Party: Sponsor-Investigator, DR. DIANE CHISESI NFS. MD. PHD., USCMDR Diane Chisesi P.I. Eng. NFS. MD. PhD., Paradyne Networks A Foundation
Organization: Paradyne Networks A Foundation (Other)
Other Study IDs: 1,20,NAS BP-B-09; CO4.588.839.500 (Other: NIH 2015 Mesh); 11063 (Other Grant/Funding Number: IRB); IRB00000553 (Other Grant/Funding Number: IRB); IORG0000432 (Other Grant/Funding Number: OHRP/FDA)
Record Dates: First submitted 2015-03-20; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Breast Cancer; Tumor; Muscle Neoplasms; Chronic Pain
Keywords: Dose Unit; Participants; Confidence Intervals; Cmax
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Muscle Neoplasms; Chronic Pain | interventions — Anastrozole; Tamoxifen; Melphalan; Fluorouracil

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples With DNA — Diagnosis of cancer or excisional biopsy for lesion not clearly benign based on previous biopsy or clinical, radiographic.
  If non-invasive cancer, incidental discovery of breast cancer on prophylactic mastectomy, incidental discovery of breast cancer on reduction mammoplasty, pre-operative biopsy proven lymph node (LN) metastases, inflammatory carcinoma, stage 3 locally advanced cancer, recurrent invasive breast cancer, or male or female diagnosed breast cancer.
  Excision of cyst, fibroadenoma, or other benign or malignant tumor. Aberrant breast tissue, duct lesion, nipple, areolar lesion, open, male, female, 1 or more lesions. Preoperative placement radiological marker, open; single lesion Each additional lesion separately identified by a preoperative radiological marker.
  Neoplasms, benign uncertain behavior,Imaging abnormalities.
  High risk lesions include but not limited to any lesion atypia or lobular carcinoma in situ.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Method(s)1/PIF Used to Evaluate: Competency Areas- Surgical care to patients with complex or recurrent neoplasms, including diagnosis and management of rare or unusual tumors.
  Determining disease stage/treatment options for individual cancer patients at time of diagnosis and throughout the disease course.
  Provide surgical care to patients with complex or recurrent neoplasms, including selecting for surgical therapy in combination with other forms of cancer treatment.
  Performing palliative surgical.
  Intervention(s): Use "Attribution", assign category code of attribution Codes: 1-5, Descriptor, Unrelated, Unlikely, Possible, Probable, Definite.
  Definitions: Use list of Adverse Events.
  Dose Units -1 mg, anastrozole. 20 mgs NOLVADEX administer to patient. Tamoxifen citrate was added to melphalan (Lphenylalanine mustard (P) and fluorouracil (F)).
  Interventions: Drug: Method(s)1 Attribution; Drug: Method(s)2 Attribution,
- Method(s)2/PIF Used to Evaluate: Competency Areas- Biologic, pharmacologic, and physiologic rationale for each form of therapy, indications, risks, and benefits of regional and systemic therapy in adjuvant and advanced disease settings.
  Nonsurgical cancer treatment modalities, including radiotherapy, chemotherapy, immunotherapy, and endocrine therapy.
  Nonsurgical palliative treatments.
  Rehabilitative services, including reconstructive surgery and physical rehabilitation.
  Tumor biology, carcinogenesis, epidemiology, tumor markers, and tumor pathology.
  Intervention(s): "Attribution" defines the relationship between the adverse event and the investigational agent(s)/intervention. Assign category code of attribution Codes: 1-5, Descriptor, Unrelated, Unlikely, Possible, Probable, Definite.
  Definitions: Use list of Adverse Events.
  Dose Units- adjuvant cytotoxic chemotherapy, added to lequo, low-dose cyclophosphamide methotrexate and fluoruracil
  Interventions: Drug: Method(s)1 Attribution; Drug: Method(s)2 Attribution,

INTERVENTIONS:
Drug: Method(s)1 Attribution — Intervention(s): "Attribution" defines the relationship between the adverse event and the investigational agent(s)/intervention. Assign the appropriate category code of attribution Codes: 1-5, Descriptor, Unrelated, Unlikely, Possible, Probable, Definite.
  Definitions: Use the Adverse Event Dose Units- Indicate the dosing units (e.g., mg) administered to the patient. TAC, Reporting Group: Participants with Disease, Description: Presence of Disease as Defined by positive reference test.
  Dosage Form: 1mg Anastrozole, given once daily. 20 mg NOLVADEX (tamoxifen citrate) tablet given once daily, (the 20 mg NOLVADEX (tamoxifen citrate) tablet is bioequivalent to the 10 mg NOLVADEX. (tamoxifen citrate) tablets.)
  Other Names: anastrazole
Drug: Method(s)2 Attribution, — Intervention(s): -"Attribution" defines the relationship between the adverse event and the investigational agent(s)/intervention. Assign the appropriate category code of attribution Codes: 1-5, Descriptor, Unrelated, Unlikely, Possible, Probable, Definite.
  Definitions: Use Adverse Events. Dose Units- Indicate the dosing units (e.g., mg) administered to the patient TAC. Reporting Group: Participant without Disease, Description: Absence of Disease as defined by negative reference test.
  Dosage Form: 1mg Anastrozole, given once daily. 20 mg NOLVADEX (tamoxifen citrate) tablet given once daily, (the 20 mg NOLVADEX (tamoxifen citrate) tablet is bioequivalent to the 10 mg NOLVADEX. (tamoxifen citrate) tablets.)
  Other Names: Tamoxifen Citrate; NOLVADEX; L phenylalanine mustard (P); Fluorouracil (f)

SUMMARY:
At a median follow-up of 33 months, the combination of anastrozole and NOLVADEX (tamoxifen citrate) did not demonstrate any efficacy benefit when compared to NOLVADEX (tamoxifen citrate) therapy given alone in all patients as well as in the hormone receptor positive subpopulation. This treatment arm was discontinued from the trial.

This study is now a combination therapy whereas the median duration of adjuvant treatment for safety evaluation is 59.8 months and 59.6 months for patients receiving anastrozole 1 mg and NOLVADEX (tamoxifen citrate) 20 mg, respectively.

DETAILED DESCRIPTION:
Of importance: (Special group- node positive disease and node negative disease).

Among 29,441 patients with ER positive or unknown breast cancer, 58% were entered into trials comparing NOLVADEX (tamoxifen citrate) to no adjuvant therapy and 42% were entered into trials comparing NOLVADEX (tamoxifen citrate) in combination with chemotherapy vs. the same chemotherapy alone. Among these patients, 54% had node positive disease and 46% had node negative disease.

The Early Breast Cancer Trialists' Collaborative Group (EBCTCG) conducted worldwide overviews of systemic adjuvant therapy for early breast cancer in 1985, 1990, and again in 1995. In 1998, 10-year outcome data were reported for 36,689 women in 55 randomized trials of adjuvant NOLVADEX (tamoxifen citrate) using doses of 20-40 mg/day for 1-5+ years. Twenty-five percent of patients received 1 year or less of trial treatment, 52% received 2 years, and 23% received about 5 years.

Forty-eight percent of tumors were estrogen receptor (ER) positive ( > 10 fmol/mg), 21% were ER poor ( < 10 fmol/l), and 31% were ER unknown.

This following study is for an alternate treatment plan. Dose specific.

ELIGIBILITY:
Inclusion Criteria:

* The Median Duration of Adjuvant Treatment for 59.8 Months and 59.6 Months for Patients Receiving Anastrozole 1 mg and NOLVADEX (Tamoxifen Citrate) 20 mg.
* Construct Patient Historical Background
* Palliative
* Pediatric- Under 2 Years of Age, 2-18 Years of Age (does unit adjustments )FYI
* Interventional Procedures
* BMD Bone Mineral Density (Data if Obtainable)
* Notate Receptor Levels (Only Women With Both Estrogen and Progesterone
* Levels 10 mo Fmol or Greater)
* Notate Radiation Therapy 6 Months (Male, Prostate Cancer, or SAST, Salvage Androgen Suppression)
* Notate Did Not Utilize Androgen Suppression as Adjunct Therapy to Radiation Therapy, Yes or no.
* Androgen Independent Prostate Cancer
* In addition: (for chronic, non-cancer pain), prescribers should determine whether the patient improves functionally on opioids, which could include an opioid trial, and whether the pain relief improves his/her ability to comply with the overall pain management program.
* Chronic Pain (Benign) Inpatient/Outpatient
* Cancer Pain
* Acute Pain, Inpatient/Outpatient
* Add here: if prudent-2.2.3.8.1.1. Dose Modification (Change)
* Has this patient received either a dose escalation or a de-escalation of this investigational agent during this course of therapy? Use the following codes:
* 1 = Yes, planned (i.e., the dose was changed according to protocol guidelines)
* 2 = Yes, unplanned (i.e., the dose change was not a part of protocol guide-lines)
* 3 = No
* 9 = Unknown
* Note: If the patient has received a previous escalation or de-escalation of this investigational agent and there has been no further change to the dose during this course, answer no.
* Construct a Least Squares Linear Regression Standard Curve, Construct a Least Squares Linear Regression, Peak Height ,
* Using data from the control (0 ppb) and fortified tissue samples, construct a least squares linear regression standard curve by plotting fortified tissue concentration against peak height (average from duplicate dose can include injection if drug is developed into injector, currently use of tablets) for the resulting equation, y = mx -t- b.

  * x = concentration (ppb) of results from chemicals or tissue from prior surgeries (if any or in progress for sample tissue)
  * y = tamoxifen citrate was added to melphalan [L-phenylalanine mustard (P) and fluorouracil (f) peak height (average value from duplicate does). This will assist in further studies for set up for adjutant cytotoxic chemotherapy if applicable.
  * m = slope
  * b = y-intercept
* Healthy volunteers/yes
* Will accept women 59-70 for use of combination drug-(both estrogen and progesterone receptor levels).

Exclusion Criteria:

* At a median follow-up of 33 months, the combination of anastrozole and NOLVADEX (tamoxifen citrate) did not demonstrate any efficacy benefit when compared to NOLVADEX (tamoxifen citrate) therapy given alone in all patients as well as in the hormone receptor positive sub-population. This treatment arm was discontinued from the trial.

Ages: 44 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In the anastrozole adjuvant trial, co-administration of anastrozole 1mg, and (tamoxifen citrate) tablets given twice a day vs. a 20 mg NOLVADEX , In cytosols derived from human breast adenocarcinomas, tamoxifen competes with estradiol for estrogen receptor protein, absorption and distribution. After initiation of therapy, steady state concentrations for tamoxifen are achieved in about 4 weeks and steady-state concentrations for N-desmethyl tamoxifen are achieved in about 8 weeks, suggesting a half-life of approximately 14 days for this metabolite.
  For this Study population-Suggest: The median duration of adjuvant treatment for safety evaluation is 59.8 months and 59.6 months for patients receiving start dose anastrozole 1 mg and NOLVADEX (tamoxifen citrate) 20 mg, respectively.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The combination of anastrozole and NOLVADEX (tamoxifen citrate)was added to adjunct cytotoxic chemothrapy | At a median follow-up of 33 months
  Among women with ER positive or unknown breast cancer and positive nodes who received about 5 years of treatment, overall survival at 10 years was 61.4% for NOLVADEX (tamoxifen citrate) vs. 50.5% for control (logrank 2p < 0.00001).
  The recurrence-free rate at 10 years was 59.7% for NOLVADEX (tamoxifen citrate) vs. 44.5% for control (logrank 2p < 0.00001). Among women with ER positive or unknown breast cancer and negative nodes who received about 5 years of treatment, overall survival at 10 years was 78.9% for NOLVADEX (tamoxifen citrate) vs. 73.3% for control (logrank 2p < 0.00001). The recurrence-free rate at 10 years was 79.2% for NOLVADEX (tamoxifen citrate) versus 64.3% for control (logrank 2p < 0.00001)
female, effective clinical care | 33 months
  Breast Cancer Resection Pathology Reporting: pT Category (Primary Tumor) and pN Category (Regional Lymph Nodes) with Histologic Grade: Percentage of breast cancer resection pathology reports that include the pT category (primary tumor), the pN category (regional lymph nodes), and the histologic grade
female, effective clinical care | 12-month
  Receptor/Progesterone Receptor (ER/PR) Positive Breast Cancer: Percentage of female patients aged 18 years and older with Stage IC through IIIC, ER or PR positive breast cancer who were prescribed tamoxifen or aromatase inhibitor (AI) during the 12-month reporting period
  *Although there a newer version of this measure is available (CMS140v2), a substantive error was discovered in the June 2013 version of this electronically specified clinical quality measure. The PQRS will require the use of the prior, December 2012 version of this measure, which is CMS140v1.

OTHER OUTCOMES:
male. effective clinical care | 6 months
  Prostate Cancer: Adjuvant Hormonal Therapy for High Risk Prostate Cancer Patients: Percentage of patients, regardless of age, with a diagnosis of prostate Cancer at high risk of recurrence receiving external beam radiotherapy to the prostate who were prescribed adjuvant hormonal therapy (GnRH agonist or antagonist

CONTACTS AND LOCATIONS:
Overall Officials: USCMDR Diane Chisesi, MD PhD CI, Principal Investigator — Chisesi, Diane M,: Army/Air Force/Mil/DHS/Other
Locations (1):
- PNAF Medical, Colorado Springs, Colorado, United States

REFERENCES:
- [Result] Anastrozole Adjuvant Trial - Study of Anastrozole compared to NOLVADEX (tamoxifen citrate) for Adjuvant Treatment of Early Breast Cancer (see CLINICAL PHARMACOLOGY - Clinical Studies) and Malignant Joint Tumor.
- [Result] Ductal Carcinoma in Situ (DCIS) The type and frequency of adverse events in the NSABP B-24 trial was consistent with those observed in the other adjuvant trials conducted with NOLVADEX (tamoxifen citrate)
- [Result] Ductal Carcinoma in Situ NSABP B-24, a double-blind, randomized trial included women with ductal carcinoma in situ (DCIS). This trial compared the addition of NOLVADEX (tamoxifen citrate) or placebo to treatment with lumpectomy and radiation therapy for women with DCIS. The primary objective was to determine whether 5 years of NOLVADEX (tamoxifen citrate) therapy (20 mg/day) would reduce the incidence of invasive breast cancer in the ipsilateral (the same) or contralateral (the opposite) breast.
- See also: Anastrozole, Chemical notes and resources, clinicaltrials.gov — https://druginfo.nlm.nih.gov/drugportal/name/anastrozole
- See also: ChemIDplus Advanced, Anastrozole — https://chem.nlm.nih.gov
- See also: ToxNet data in PubChem — https://pubchemdocs.ncbi.nlm.nih.gov/about